CLINICAL TRIAL: NCT05838651
Title: The Combination of BioHorizon's Striate+ Membrane in Conjunction With MinerOss X Plug for Providing Hard Tissue Regeneration in Socket Preservation Procedure
Brief Title: Socket Preservation With BioHorizon's Striate+ Membrane and MinerOss X Plug
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Dental Medicine (Other)
Collaborators: Camlog Oral Reconstruction Foundation (Other); BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Chia-Yu Chen, Assistant Professor, Department of Oral Medicine, Infection, and Immunity, Harvard School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0179
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Socket Preservation
Keywords: Bone Graft; Membrane; Extraction

STUDY DESIGN:
Intervention Model Description: Randomized Control Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bone Graft Alone (Active Comparator): Socket preservation sites with bone graft (MinerOss® X Plug) alone without complete flap closure (secondary intention healing) (n=10)
  Interventions: Device: MinerOss® X Plug
- Bone Graft + Membrane (Experimental): Socket preservation sites with bone graft (MinerOss® X Plug) and a non-crosslinked collagen membrane without complete flap closure (secondary intention healing) (n=10)
  Interventions: Device: MinerOss® X Plug; Device: Striate+ Membrane

INTERVENTIONS:
Device: MinerOss® X Plug — A xenograft composed of 80% bovine cancellous particulate and 20% bovine Type I collagen.
Device: Striate+ Membrane — A non-crosslinked collagen covering used to keep bacteria out and hold the bone graft in place.
  Arms: Bone Graft + Membrane

SUMMARY:
The primary objective of this proposed clinical trial is to provide detailed comparison and evidence of new bone formation in patients undergoing socket preservation utilizing MinerOss® X Plug with and without Striate+ Membrane to maintain ridge dimension after a tooth extraction.

DETAILED DESCRIPTION:
The primary objective of this proposed clinical trial is to provide detailed comparison and evidence of new bone formation in patients undergoing socket preservation utilizing two widely accepted treatment modalities that are used to maintain ridge dimension after a tooth extraction.

The specific aims of the study are:

1. To demonstrate the efficacy of a Striate+ membrane in conjunction with a bone graft substitute for providing hard tissue regeneration in the socket preservation procedure.
2. To determine the safety of Striate+ membrane when primary flap closure over the membrane is not achieved in the socket preservation procedure.
3. To provide detailed evidence of new bone formation in patients undergoing socket preservation procedures by means of clinical, radiographic, histologic, and histomorphometric analyses.

It is currently unclear if one treatment is more effective than the other. The two treatments being compared are:

Treatment 1: Socket preservation sites with bone graft (MinerOss® X Plug) alone without complete flap closure (secondary intention healing) (n=10) Treatment 2: Socket preservation sites with bone graft (MinerOss® X Plug) and a non-crosslinked collagen membrane without complete flap closure (secondary intention healing) (n=10)

MinerOss® X Plug: A xenograft composed of 80% bovine cancellous particulate and 20% bovine Type I collagen. The 20% collagen prevents particulate migration.

Striate+ Membrane: A non-crosslinked collagen covering used to keep bacteria out and hold the bone graft in place.

Secondary intention healing (without complete flap closure): The wound edges are not brought together (i.e. knee scrape).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 20-70 years of age, who requests dental implant treatment option for rehabilitation.
* Subjects who are willing to sign an informed consent, participate and return for follow-up visits.
* Subjects without significant medical history and currently not on medications that might complicate our results.
* Has a single-rooted tooth (upper and lower premolars to premolars) requiring extraction with two neighboring teeth on either side of it and intact bony walls.

Exclusion Criteria:

* Subjects who do not meet all the inclusion criteria or who will not cooperate with the protocol schedule.
* Subjects who received and failed a previously placed dental implant.
* Subjects who require additional ridge augmentation procedure in the area to achieve adequate bone volume for the placement of dental implants.
* Subjects who have significant untreated periodontal disease, caries, infection or chronic inflammation in the oral cavity within two adjacent tooth positions of the clinical trial area.
* Subjects who have used nicotine-containing products within 3 weeks prior to surgery.
* Subjects who are insulin-dependent diabetic or if their Hgb1c levels > 6.5%.
* Subjects who have had a history of malignancy within the past 5 years (except for basal or squamous cell carcinoma of the skin or in situ cervical carcinoma).
* Subjects who are nursing or pregnant.
* Subjects who are presently taking medications (except estrogen/progesterone therapy) or those who are undergoing treatment that in known to have an effect on bone turnover.
* Subjects who have diseases that affect bone metabolism (excluding idiopathic osteoporosis).
* Subjects with a history of an autoimmune disease, documented allergy or multiple allergies to any component of the agents used in this study.
* Difficult extraction with potential disruption / fracture of the alveolar bone.
* Acutely infected defect site.
* Subjects who are presently taking blood thinner medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
radiographic ridge width | 12 months
  To provide detailed evidence of new bone formation in patients undergoing socket preservation procedures.

SECONDARY OUTCOMES:
gingival thickness | 12 months
  To assess soft tissue changes.
radiographic alveolar height | 12 months
  To assess radiographic hard tissue changes.
clinical alveolar height and width | 12 months
  To assess clinical hard tissue changes.

CONTACTS AND LOCATIONS:
Overall Officials: David M Kim, DDS, DMSc, Principal Investigator — Harvard School of Dental Medicine
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05838651/ICF_000.pdf